CLINICAL TRIAL: NCT02506959
Title: Panobinostat Combined With High-Dose Gemcitabine/Busulfan/Melphalan With Autologous Stem Cell Transplant for Patients With Refractory/Relapsed Myeloma
Brief Title: Panobinostat, Gemcitabine Hydrochloride, Busulfan, and Melphalan Before Stem Cell Transplant in Treating Patients With Refractory or Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0516; NCI-2015-01308 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0516 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Plasma Cell Leukemia; Plasmacytoma; Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Leukemia, Plasma Cell; Plasmacytoma; Multiple Myeloma | interventions — Busulfan; Gemcitabine; Melphalan; Panobinostat; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1_1st Auto TP Conditioned with panobinostat and Gem/Bu/Mel (Experimental): Patients receive panobinostat PO QD on days -9 to -2, gemcitabine hydrochloride IV over 4 hours on days -8 and -3, busulfan IV over 3 hours on days -8 to -5, and melphalan IV over 30 minutes on days -3 and -2. Patients then undergo autologous peripheral blood stem cell transplant on day 0.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Busulfan; Drug: Gemcitabine Hydrochloride; Drug: Melphalan; Drug: Panobinostat; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Pharmacological Study
- Cohort 2_2nd Auto TP Conditioned with panobinostat and Gem/Bu/Mel (Experimental): Patients receive panobinostat PO QD on days -9 to -2, gemcitabine hydrochloride IV over 4 hours on days -8 and -3, busulfan IV over 3 hours on days -8 to -5, and melphalan IV over 30 minutes on days -3 and -2. Patients then undergo autologous peripheral blood stem cell transplant on day 0.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Busulfan; Drug: Gemcitabine Hydrochloride; Drug: Melphalan; Drug: Panobinostat; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Pharmacological Study

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous peripheral blood stem cell transplant
  Other Names: Autologous Hematopoietic Cell Transplantation
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; FF 10832; FF-10832; FF10832; Gemcitabine HCI; Gemzar; LY-188011; LY188011
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Panobinostat — Given PO
  Other Names: Faridak; LBH589
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo autologous peripheral blood stem cell transplant
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood; Peripheral Blood Progenitor Cell Transplantation; PERIPHERAL BLOOD STEM CELL TRANSPLANT; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well panobinostat, gemcitabine hydrochloride, busulfan, and melphalan before stem cell transplant work in treating patients with multiple myeloma that does not respond to treatment (refractory) or has returned (relapsed). Panobinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving high-dose chemotherapy, such as gemcitabine hydrochloride, busulfan, and melphalan, before a peripheral blood stem cell transplant helps kill any cancer cells that are in the body and helps make room in the patient's bone marrow for new blood-forming cells (stem cells) to grow. Previously collected stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the progression-free survival (PFS) in patients with refractory or relapsed myeloma receiving panobinostat/gemcitabine hydrochloride (gemcitabine)/busulfan/melphalan (panobinostat/Gem/Bu/Mel) with autologous stem-cell transplant, either as a first or a salvage stem-cell transplant.

SECONDARY OBJECTIVES:

I. To evaluate the complete response (CR) rate. II. To determine the overall survival (OS). III. To determine the CR + very good partial remission (VGPR) rate. IV. To determine the overall response rate (ORR). V. To determine minimal residual disease posttransplant, measured by multiparametric flow cytometry (MFC).

VI. To describe the toxicity profile of panobinostat/Gem/Bu/Mel. VII. To analyze the predictive value of pretransplant levels in myeloma cells of X-box binding protein 1 (XBP1), inositol-requiring enzyme 1 (IRE1), unspliced XBP1 (XBP1u), sliced XBP1 (XPB1s), XBP1u/XPBs ratio and v-myc myelocytomatosis viral oncogene homolog (avian) (Myc), by analyzing their correlation with CR, VGPR+CR and response rate (RR).

VIII. To study the prognostic effect of pretransplant levels in myeloma cells of XBP1, IRE1, XBP1u, XPB1s, XBP1u/XPBs ratio and Myc, by analyzing their correlation with PFS and OS.

OUTLINE:

Patients receive panobinostat orally (PO) once daily (QD) on days -9 to -2, gemcitabine hydrochloride intravenously (IV) over 4 hours on days -8 and -3, busulfan IV over 3 hours on days -8 to -5, and melphalan IV over 30 minutes on days -3 and -2. Patients then undergo autologous peripheral blood stem cell transplant on day 0.

After completion of study treatment, patients are followed up at 1 month, 100 days, 6 months, 1 year, and then every 3-6 months for at least 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Refractory or relapsed myeloma, defined as one or more of the following:

  * Treated with first-line therapy including at least 2 cycles of lenalidomide, bortezomib or thalidomide, and one or more of the following:

    * Less than partial response (PR) to first-line therapy
    * Relapse after first (1st) line therapy
  * High-risk cytogenetics, defined by deletion (del)(13q) by conventional cytogenetics, or by del(17p), t(4;14), t(14;16), t(14;20) or 1q+ by fluorescence in situ hybridization (FISH)
  * Relapse after a prior autologous stem cell transplant (ASCT)
  * Plasma cell leukemia
  * Soft tissue plasmacytoma
* Serum creatinine =< 1.8 mg/dL and/or estimated serum creatinine clearance >= 50 ml/min
* Serum glutamic oxaloacetic transaminase (SGOT) and/or serum glutamate pyruvate transaminase (SGPT) =< 3 x upper limit of normal
* Serum bilirubin =< 2 x upper limit of normal, unless proven to be due to disease involvement
* Alkaline phosphatase =< 2 x upper limit of normal, unless proven to be due to disease involvement
* Adequate pulmonary function with forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and diffusion capacity of the lung for carbon monoxide (DLCO) >= 50% of expected corrected for hemoglobin and/or volume
* Adequate cardiac function with left ventricular ejection fraction >= 40%
* No uncontrolled arrhythmias or symptomatic cardiac disease
* Clinically euthyroid; note: patients are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism
* Zubrod performance status < 2
* Negative beta-human chorionic gonadotropin (HCG) test in a woman of child-bearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization
* Availability of >= 2.5 million cluster of differentiation (CD)34+ cells/kg previously apheresed
* Ability to provide written informed consent

Exclusion Criteria:

* Prior whole brain irradiation
* Having received radiation therapy to head and neck (excluding eyes), and internal organs of chest, abdomen or pelvis in the month prior to enrollment
* Active hepatitis B, either active carrier (hepatitis B surface antigen positive [HBsAg +]) or viremic (hepatitis B virus [HBV] deoxyribonucleic acid [DNA] >= 10,000 copies/mL, or >= 2,000 IU/mL)
* Evidence of either cirrhosis or stage 3-4 liver fibrosis in patients with chronic hepatitis C or positive hepatitis C serology
* Active infection requiring parenteral antibiotics
* Known positivity for human immunodeficiency virus (HIV)
* Autologous stem-cell transplant in the previous six months
* Needing valproic acid for any medical condition during the study or within 5 days prior to first panobinostat treatment
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of panobinostat
* Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes or active or uncontrolled infection) including abnormal laboratory values, that could cause unacceptable safety risks or compromise compliance with the protocol
* Impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

  * History or presence of sustained ventricular tachyarrhythmia; (patients with a history of atrial arrhythmia are eligible but should be discussed with Secura Bio, Inc (Secura Bio) prior to enrollment)
  * Any history of ventricular fibrillation or torsade de pointes
  * Bradycardia defined as heart rate (HR) < 50 beats per minute (bpm); patients with pacemakers are eligible if HR >= 50 bpm
  * Screening electrocardiogram (ECG) with a corrected QT (QTc) > 470 msec
  * Right bundle branch block + left anterior hemiblock (bifascicular block)
  * Myocardial infarction or unstable angina =< 12 months prior to starting study drug
  * Other clinically significant heart disease (e.g., congestive heart failure [CHF] New York [NY] Heart Association class III or IV , uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
* Have undergone major surgery =< 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Prior malignancy with in the last 5 years (except for basal or squamous cell carcinoma, or in situ cancer of the cervix)
* Any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff
* Received targeted agents within 2 weeks or within 5 half-lives of the agent and active metabolites (whichever is longer) and who have not recovered from side effects of those therapies
* Having received immunotherapy or chemotherapy within 2 weeks; or radiation therapy to > 30% of marrow-bearing bone within =< 2 weeks prior to starting study treatment; or who have not yet recovered from side effects of such therapies
* Grade >= 3 nonhematological toxicity from prior therapy that has not resolved to =< grade 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yago L Nieto, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1_1st Auto TP Conditioned With Panobinostat and Gem/Bu/Mel; Cohort 2_2nd Auto TP Conditioned With Panobinostat and Gem/Bu/Mel: Patients receive panobinostat PO QD on days -9 to -2, gemcitabine hydrochloride IV over 4 hours on days -8 and -3, busulfan IV over 3 hours on days -8 to -5, and melphalan IV over 30 minutes on days -3 and -2. Patients then undergo autologous peripheral blood stem cell transplant on day 0.
  Autologous Hematopoietic Stem Cell Transplantation: Undergo autologous peripheral blood stem cell transplant
  Busulfan: Given IV
  Gemcitabine Hydrochloride: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Melphalan: Given IV
  Panobinostat: Given PO
  Peripheral Blood Stem Cell Transplantation: Undergo autologous peripheral blood stem cell transplant
  Pharmacological Study: Correlative studies
Period: Overall Study
Arm/Group | Cohort 1_1st Auto TP Conditioned With Panobinostat and Gem/Bu/Mel | Cohort 2_2nd Auto TP Conditioned With Panobinostat and Gem/Bu/Mel
Started | 50 | 33
Completed | 48 | 32
Not Completed | 2 | 1
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1_1st Auto TP Conditioned With Panobinostat and Gem/Bu/Mel | Cohort 2_2nd Auto TP Conditioned With Panobinostat and Gem/Bu/Mel | Total
Number analyzed (Participants) | 50 | 33 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 33 | 81
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 35 | 18 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 2 | 11
  Not Hispanic or Latino | 41 | 31 | 72
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 33 | 83

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Number of participants alive and disease free one year post auto transplant in patients with refractory or relapsed myeloma receiving panobinostat/gemcitabine/busulfan/melphalan (panobinostat/Gem/Bu/Mel) with autologous stem-cell transplant, either as a first or a salvage stem-cell transplant.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1_1st Auto TP Conditioned With Panobinostat and Gem/Bu/Mel | Cohort 2_2nd Auto TP Conditioned With Panobinostat and Gem/Bu/Mel
Number analyzed (Participants) | 50 | 33
Participants | 38 | 24

2. Secondary Outcome: Overall Survival (OS)
Description: Number of participants with refractory or relapse Myeloma who still remain alive two years post transplant
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1_1st Auto TP Conditioned With Panobinostat and Gem/Bu/Mel | Cohort 2_2nd Auto TP Conditioned With Panobinostat and Gem/Bu/Mel
Number analyzed (Participants) | 50 | 33
Participants | 27 | 16

3. Secondary Outcome: Participants Who Experienced Grade 3 or Higher Adverse Events
Description: Number of Participants who experienced grade 3 or higher Adverse Events during the first 100 days of the transplant.
Time Frame: Up to day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1_1st Auto TP Conditioned With Panobinostat and Gem/Bu/Mel | Cohort 2_2nd Auto TP Conditioned With Panobinostat and Gem/Bu/Mel
Number analyzed (Participants) | 50 | 33
Participants | 47 | 29

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Cohort 1_1st Auto TP Conditioned With Panobinostat and Gem/Bu/Mel | Cohort 2_2nd Auto TP Conditioned With Panobinostat and Gem/Bu/Mel
All-Cause Mortality (participants affected / at risk) | 23/50 | 17/33
Serious Adverse Events (participants affected / at risk) | 2/50 | 4/33
Other Adverse Events (participants affected / at risk) | 47/50 | 30/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1_1st Auto TP Conditioned With Panobinostat and Gem/Bu/Mel (N=50) | Cohort 2_2nd Auto TP Conditioned With Panobinostat and Gem/Bu/Mel (N=33)
AST increased (Investigations) | 0 (0) | 1 (1)
Bleeding (no GI no PUL) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
DAH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Fungal (Infections and infestations) | 1 (1) | 2 (2)
Oral mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
T bilirubin increased (Investigations) | 0 (0) | 1 (1)
Viral (Infections and infestations) | 1 (1) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1_1st Auto TP Conditioned With Panobinostat and Gem/Bu/Mel (N=50) | Cohort 2_2nd Auto TP Conditioned With Panobinostat and Gem/Bu/Mel (N=33)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
ALK increased (Investigations) | 2 (2) | 3 (3)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (1)
ALT increased (Investigations) | 25 (25) | 20 (20)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
AST increased (Investigations) | 10 (10) | 6 (6)
Bacterial (Infections and infestations) | 18 (18) | 14 (14)
Bleeding (no GI no PUL) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
CD OTH (Cardiac disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 7 (7) | 6 (6)
Diarrhea (General disorders) | 43 (43) | 28 (28)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dysgeusia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysrhythmia (Cardiac disorders) | 10 (10) | 7 (7)
Ejection fraction decreased (Cardiac disorders) | 1 (1) | 1 (1)
Engraftment syndrome (Immune system disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 43 (43) | 28 (28)
Fever (General disorders) | 11 (11) | 7 (7)
Fluid overload (General disorders) | 36 (36) | 25 (25)
Fungal (Infections and infestations) | 3 (3) | 2 (2)
GI OTH (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 3 (3)
Hemorrhagic Cystitis (Renal and urinary disorders) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 10 (10) | 9 (9)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 46 (46) | 30 (30)
NE OTH (Nervous system disorders) | 1 (1) | 0 (0)
NE VIS (Nervous system disorders) | 1 (1) | 1 (1)
Oral mucositis (Gastrointestinal disorders) | 47 (47) | 26 (26)
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 8 (8) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 27 (27) | 23 (23)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
T bilirubin increased (Investigations) | 15 (15) | 12 (12)
Thromboembolic event (Vascular disorders) | 3 (3) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Viral (Infections and infestations) | 18 (18) | 23 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT02506959/Prot_SAP_000.pdf